CLINICAL TRIAL: NCT07154433
Title: Effect of a Postoperative Multimodal Analgesic Protocol Predominantly Based on Non-Opioid Medications vs Opioid-Based Analgesia on Pain After Minimally Invasive Ankle Surgery: A Noninferiority Randomized Clinical Trial
Brief Title: A Study on Reducing Opioid Use After Minimally Invasive Ankle Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-0286
Record Dates: First submitted 2025-07-10; First posted 2025-09-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Ankle (Ligaments); Instability (Old Injury); Ankle Sprain; Talus Osteochondral Defect; Opioid Analgesia; Non-Opioid Pain Management
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: This interventional study employs a parallel - group, randomized, assessor - blinded design to compare the effectiveness and safety of non - opioid versus opioid medications for perioperative analgesia in ankle arthroscopy patients.
  Randomization: Eligible participants (n = 110) are randomly assigned in a 1:1 ratio to either the non - opioid or opioid group using a computer - generated random number sequence. The randomization process is conducted by an independent statistician, ensuring unbiased allocation and minimizing selection bias.
  Interventions:
  Non - opioid group: Receives a multimodal non - opioid analgesic regimen, including celecoxib and acetaminophen, aiming to reduce opioid exposure and associated risks such as addiction, respiratory depression, and gastrointestinal adverse events.
  Opioid group: Administered an opioid - based regimen with oxycodone - acetaminophen, representing the standard clinical practice for postoperative pain control.
  Blinding: To prevent assessment b
Who Masked: Investigator
Masking Description: This study employs investigator masking (also known as single - blind) to minimize bias in data collection and assessment. Eligible participants undergoing ankle arthroscopy are randomly assigned to either the non - opioid or opioid analgesia group using a computer - generated random number sequence. The randomization process is managed by an independent statistician, who assigns participants to groups and stores this information securely.
  Investigators responsible for direct patient interactions, including administering medications, assessing pain scores (Numeric Rating Scale, NRS), recording adverse events, and evaluating patient - reported outcomes (such as PROMIS questionnaires), are unaware of the participants' assigned groups. This masking approach ensures that their evaluations remain objective and are not influenced by expectations regarding the effectiveness or safety of the intervention.
  To maintain blinding integrity, study medications are packaged identically, and the label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Opioid Analgesia Group (Experimental): Participants in this group will receive a multimodal non - opioid analgesic regimen. The treatment includes celecoxib(Flurbiprofen axetil) and acetaminophen(Jingxin (a Chinese pharmaceutical company)), aiming to provide effective pain relief while reducing the use of opioids and minimizing associated risks such as addiction, respiratory depression, and gastrointestinal adverse events during the perioperative period of ankle arthroscopy.
  Interventions: Drug: Non-opioid analgesic regimen
- Opioid Analgesia Group (Active Comparator): This group will be administered an opioid - based regimen with oxycodone - acetaminophen(Parecoxib). It represents the standard clinical practice for postoperative pain control and serves as a reference to compare the efficacy and safety of the non - opioid regimen in managing pain after ankle arthroscopy.
  Interventions: Drug: Opioid Analgesic Regimen

INTERVENTIONS:
Drug: Opioid Analgesic Regimen — Participants will take 5 mg/325 mg of oxycodone - acetaminophen every 6 hours as needed for pain, with a maximum of 4 doses per day. Rescue analgesia protocol: a limited rescue prescription of oxycodone/acetaminophen (containing 5 mg oxycodone), to be taken every 2 hours as needed, with no more than 10 tablets per day, and only if adequate pain relief is not achieved (defined as NRS score ≥ 4).
  Arms: Opioid Analgesia Group
Drug: Non-opioid analgesic regimen — Immediately after surgery, patients will receive oral acetaminophen 500 mg plus celecoxib 400 mg. Thereafter, celecoxib 200 mg BID and acetaminophen 500 mg Q6H will be administered. Rescue analgesia protocol: a limited rescue prescription of oxycodone/acetaminophen (containing 5 mg oxycodone), to be taken every 2 hours as needed, with no more than 10 tablets per day, and only if adequate pain relief is not achieved (defined as NRS score ≥ 4).
  Arms: Non-Opioid Analgesia Group

SUMMARY:
Study Title Effect of a Postoperative Multimodal Analgesic Protocol Predominantly Based on Non-Opioid Medications vs Opioid-Based Analgesia on Pain After Minimally Invasive Ankle Surgery: A Noninferiority Randomized Clinical Trial

Purpose This study aims to compare the pain control effect and side effects of non-opioid versus opioid medications in patients undergoing ankle arthroscopy. The goal is to find a safer analgesic strategy to reduce opioid use and related risks (e.g., addiction, respiratory depression) while maintaining effective postoperative pain management.

Design Study Type: Prospective, randomized controlled trial. Participants: 110 adults (18-65 years) scheduled for ankle arthroscopy and Mini-open ankle surgery under general anesthesia.

Interventions:

Experimental Group: Non-opioid regimen (celecoxib + acetaminophen). Control Group: Opioid regimen (oxycodone + acetaminophen). Assessments: Pain scores (NRS) at 2 hours,6 hours,12 hours, 24 hours, and days 2-6 postoperatively; Area under the curve (AUC\_{0-24}) of Numerical Rating Scale (NRS) pain intensity scores from 0-24 hours.adverse events (e.g., nausea, constipation); The total consumption of additional rescue opioids, expressed as oral morphine equivalent dose (OME); patient satisfaction.

Key Eligibility Able to provide informed consent. ASA physical status I-II. BMI 16-32 kg/m². Exclusion criteria: Chronic pain, opioid use history, allergies to study drugs, or severe organ dysfunction.

Benefits & Risks Benefits: Standardized analgesia management and personalized pain monitoring; potential contribution to safer clinical pain protocols.

Risks: Opioids may cause nausea, sedation, or respiratory depression; non-opioids may carry risks of gastrointestinal bleeding or liver injury. Emergency support is available for severe events.

Contact Information

For more details, contact the research team at Zhejiang University Second Affiliated Hospital:

Phone: 0571-87783759 Email: keyanlunli_zheer@163.com This trial is registered to evaluate non-opioid alternatives for ankle arthroscopy pain control, prioritizing patient safety and evidence-based care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old. Scheduled for elective ankle arthroscopy under general anesthesia. American Society of Anesthesiologists (ASA) physical status I or II. Body mass index (BMI) 16-32 kg/m². Able to understand and sign the informed consent form. Willing and able to comply with study procedures, including follow - up visits and outcome assessments.

Exclusion Criteria:

* History of chronic pain (pain lasting >3 months) or current use of opioid medications within the past 3 months.

Known allergies or contraindications to study medications (celecoxib, acetaminophen, oxycodone, tramadol, dezocine).

Severe cardiovascular, hepatic, renal, or respiratory dysfunction (ASA ≥ III). History of substance abuse, alcohol dependence, or significant psychiatric disorders.

Pregnant or breastfeeding women. Participation in another clinical trial within the past 30 days. Unstable medical conditions that may interfere with study participation or outcome assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain score at 24 hours post-operation | 24 hours after ankle arthroscopy
  The pain score will be assessed using the Numeric Rating Scale (NRS), where 0 represents "no pain" and 10 represents "the worst pain imaginable." This score reflects the patient's subjective experience of pain intensity 24 hours after ankle arthroscopy. By comparing the NRS scores between the non - opioid analgesia group and the opioid analgesia group, we can evaluate the effectiveness of each intervention in managing acute postoperative pain.

SECONDARY OUTCOMES:
Area under the curve (AUC_{0-24}) of Numerical Rating Scale (NRS) pain intensity scores from 0-24 hours. | Within 24 hours postoperatively
  The area under the curve (AUC) of NRS pain scores within the first 24 hours will be calculated using NRS measurements at 2, 6, 12, and 24 hours postoperatively, providing an accurate estimate of the patient's overall pain experience during the 24-hour period.
The total consumption of additional rescue opioids, expressed as oral morphine equivalent dose (OME) | From immediately after surgery until 6 days post - operation
  This indicator reflects whether pain control in the non-opioid group is adequate. If pain control is insufficient, patients will consume more opioids for rescue, thereby allowing an inference on the analgesic efficacy of the non-opioid regimen.
Incidence of adverse events | From the start of medication administration until 6 days post - operation
  Adverse events related to the analgesic regimens will be recorded, including but not limited to nausea, vomiting, constipation, dizziness, sedation, respiratory depression, and gastrointestinal bleeding. The occurrence rate of each adverse event will be calculated for both groups to evaluate the safety profiles of the non - opioid and opioid interventions.
Patient - reported satisfaction | 6 days post - operation
  Participants will complete a 4-point likert scale to describe his satisfaction of the pain manegement at 6 days post - operation. The questionnaire assesses patients' overall satisfaction with the pain management strategy, including aspects such as effectiveness of pain relief, tolerability of medications, and impact on daily activities. Scores range from 1 (extremely dissatisfied) to 4 (extremely satisfied).
Patient - reported outcome measures (PROMIS) scores | Baseline (pre - operation), and 6 days post - operation
  Participants will fill out the PROMIS Pain Interference - Short Form (PI - SF) . it evaluate the impact of pain on daily function , respectively. Scores are standardized, with higher values indicating greater interference or disturbance.
Pain score on the second postoperative day | 2 hours post - operation; 2 - 6 days post - operation
  Pain intensity will be evaluated using the Numeric Rating Scale (NRS, 0 = no pain, 10 = worst pain imaginable) at second postoperative day. the scores help to comprehensively assess the time - course of pain relief provided by each intervention.
Pain score on the third postoperative day | the third postoperative day
  Pain intensity will be evaluated using the Numeric Rating Scale (NRS, 0 = no pain, 10 = worst pain imaginable) at third postoperative day. the scores help to comprehensively assess the time - course of pain relief provided by each intervention.
Pain score on the forth postoperative day | the forth postoperative day
  Pain intensity will be evaluated using the Numeric Rating Scale (NRS, 0 = no pain, 10 = worst pain imaginable) at forth postoperative day. the scores help to comprehensively assess the time - course of pain relief provided by each intervention.
Pain score on the fifth postoperative day | on the fifth postoperative day
  Pain intensity will be evaluated using the Numeric Rating Scale (NRS, 0 = no pain, 10 = worst pain imaginable) at fifth postoperative day. the scores help to comprehensively assess the time - course of pain relief provided by each intervention.
Pain score on the sixth postoperative day | the sixth postoperative day
  Pain intensity will be evaluated using the Numeric Rating Scale (NRS, 0 = no pain, 10 = worst pain imaginable) at sixth postoperative day. the scores help to comprehensively assess the time - course of pain relief provided by each intervention.
Insomnia Severity Index | Baseline (pre - operation), and 6 days post - operation
  To assess the subjective severity of insomnia before and after surgery, its impact on daytime functioning, and the degree of distress caused by sleep problems.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China